CLINICAL TRIAL: NCT00918216
Title: Spectroscopy of Breast Tissue
Status: Completed | Type: Observational
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE8107; P30CA043703 (NIH); CASE8107 (Other: Case Comprehensive Cancer Center); CASE-8107-CC441 (Other: Cancer Center IRB)
Record Dates: First submitted 2009-06-10; First posted 2009-06-11 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — In Situ Hybridization, Fluorescence; Immunohistochemistry; Spectrometry, Fluorescence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — This study will involve up to 200 female patients already undergoing needle biopsy or surgical excision of a breast lesion identified clinically.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: fluorescence in situ hybridization — Additional histochemical, immunohistochemical, and fluorescence in situ stains may be performed to support the diagnosis or to better understand the spectroscopy results.
Other: immunohistochemistry staining method — Additional histochemical, immunohistochemical, and fluorescence in situ stains may be performed to support the diagnosis or to better understand the spectroscopy results.
Other: medical chart review — Patients' medical charts are reviewed to obtain clinical information
Procedure: fluorescence spectroscopy — The freshly excised breast tissue samples are analyzed ex vivo by fluorescence, reflectance, and/or Raman spectroscopy.
Procedure: histopathologic examination — Hematoxylin and eosin stained sections of the tissue samples are examined by light microscopy for histopathological analysis.
Procedure: light-scattering spectroscopy — The freshly excised breast tissue samples are analyzed ex vivo by fluorescence, reflectance, and/or Raman spectroscopy.

SUMMARY:
RATIONALE: Diagnostic procedures, such as laser spectroscopy, may help find and diagnose breast cancer.

PURPOSE: This phase I trial is studying laser spectroscopy to see how well it works in diagnosing breast cancer in women with breast lesions.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether laser spectroscopy of breast tissue performed ex vivo can effectively distinguish between benign and malignant breast tumors in women undergoing needle biopsy or surgical excision of a breast lesion identified clinically.

OUTLINE: Patients undergo tissue sample collection via needle biopsy or surgical excision of a breast lesion. A radiogram of the sample may be obtained to identify target areas for spectroscopic evaluation. The freshly excised breast tissue samples are analyzed ex vivo by fluorescence, reflectance, and/or Raman spectroscopy. After completion of the spectroscopic examination, the tissue samples are submitted for diagnostic pathologic evaluation. Hematoxylin and eosin stained sections of the tissue samples are examined by light microscopy for histopathological analysis. The results of the pathological examination are then compared with the spectroscopic findings and radiological findings (if the biopsy was performed for a suspect lesion on mammography) to determine if any correlation can be established and which spectroscopic technique provides the most useful diagnostic information. Additional histochemical, immunohistochemical, and fluorescence in situ stains may be performed to support the diagnosis or to better understand the spectroscopy results.

Patients' medical charts are reviewed to obtain clinical information (e.g., age, sex, and race; results of pathology reports and reports of ancillary studies, including estrogen receptor, progesterone receptor, and HER-2 receptor testing, for the surgical specimen being studied and for any other related surgical specimens; menstrual status and date of last menstrual period; clinical history of breast mass or abnormal mammogram and related mammography report; clinical history of hormone replacement therapy, birth control pills, or oophorectomy; and clinical history of chemotherapy or other adjuvant therapy for breast cancer).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Clinically identified breast lesion
* Planning to undergo needle biopsy or surgical excision of the breast lesion

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will involve up to 200 female patients already undergoing needle biopsy or surgical excision of a breast lesion identified clinically. The patients will be recruited from the General Surgery and Radiology practices of the co-investigators.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2008-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Ability of laser spectroscopy performed ex vivo to effectively distinguish between benign and malignant breast tumors | At the time of biopsy
  The data will be taken with a portable spectroscopy system that can perform fluorescence, reflectance and Raman spectroscopy simultaneously through a single fiber optic probe.

CONTACTS AND LOCATIONS:
Overall Officials: Maryann Fitzmaurice, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States